CLINICAL TRIAL: NCT06690346
Title: Systematic Oral Care Education for Preventing Oral Complications in Patients Undergoing Radiotherapy for Head and Neck Malignancies: A Randomized Controlled Trial
Brief Title: Systematic Oral Education for Prevention of Oral-related Complications Caused by Radiotherapy for Head and Neck Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: West China Hospital (Other)
Responsible Party: Principal Investigator, Xingchen Peng, Study director, West China Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2024-1262
Record Dates: First submitted 2024-11-08; First posted 2024-11-15 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2025-12

CONDITIONS: Malignant Tumor of Head and/or Neck; Radiotherapy; Complications
MeSH Terms: conditions — Head and Neck Neoplasms

STUDY DESIGN:
Intervention Model Description: Intervention group: Systematic oral health education Control group: Routine oral health education
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): Systematic oral health education
  Interventions: Other: Systematic oral health education
- Control group (Other): Routine oral health education
  Interventions: Other: Routine oral health education

INTERVENTIONS:
Other: Systematic oral health education — Provide systematic oral health education to patients in experimental group, including oral hygiene instruction and dietary instruction
  Arms: Experimental group
Other: Routine oral health education — Provide routine oral health education to patients in control group, including routine oral self-care instruction
  Arms: Control group

SUMMARY:
A study on the efficacy of systematic oral health education for the prevention of oral-related complications caused by radiotherapy for head and neck malignant tumors

DETAILED DESCRIPTION:
The goal of this clinical trial is to investigate the efficacy of systematic oral health education for oral-related complications in patients with head and neck malignant tumors who receive radiotherapy. The main question it aims to answer is:

the efficacy of systematic oral health education for the prevention oral-related complications caused by radiotherapy for head and neck malignant tumors

Participants will:

be given systematic oral health education or routine oral health education be evaluated to learn the efficacy of systematic oral health education for the prevention of oral-related complications caused by radiotherapy for head and neck malignant tumors Researchers will compare systematic oral health education group with routine oral health education group to see if systematic oral health education has good efficacy for the prevention of oral-related complications caused by radiotherapy for head and neck malignant tumors.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with malignant tumors of the head and neck without metastasis
* Age ≥18, ≤80 years old
* ECOG_PS score ≤2
* Receiving radiotherapy alone or concurrent radiotherapy with a radiation dose of >50 Gy
* Signed informed consent form

Exclusion Criteria:

* Patients with oral mucositis due to allergic reactions to certain foods, medications, or oral care products
* Have a history of head and neck radiotherapy
* Poor oral hygiene or severe periodontitis
* Poor compliance
* Other patients who, in the opinion of the investigator, are not suitable for participation in this study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2024-11-26 (Actual); Primary Completion 2025-06-26 (Actual); Study Completion 2025-06-26 (Actual)

PRIMARY OUTCOMES:
The incidence of oral mucositis (OM) | 1 week before radiotherapy; weekly during radiotherapy(until 7 weeks); 1, 2, 3 months after the end of radiotherapy
  Oral mucositis is assessed by trained physicians according to World Health Organization (WHO) oral toxicity Scale(grade 1-5); Higher grade indicates more severe symptoms

SECONDARY OUTCOMES:
The incidence of severe oral mucositis (SOM) (WHO grade ≥3) | 1 week before radiotherapy; weekly during radiotherapy(until 7 weeks); 1, 2, 3 months after the end of radiotherapy
  Oral mucositis is assessed by trained physicians according to World Health Organization (WHO) oral toxicity Scale(grade 1-5); Higher grade indicates more severe symptoms
The time to onset of severe oral mucositis (SOM) (WHO grade ≥3) | 1 week before radiotherapy; weekly during radiotherapy(until 7 weeks); 1, 2, 3 months after the end of radiotherapy
  Time from the first day of radiotherapy to the first determination of SOM.
The duration of severe oral mucositis (WHO grade ≥3) | 1 week before radiotherapy; weekly during radiotherapy(until 7 weeks); 1, 2, 3 months after the end of radiotherapy
  The first determination of SOM to the first instance of non-severe OM (WHO grade <3), without a subsequent instance of SOM.
The time to onset of any-grade oral mucositis (OM) | 1 week before radiotherapy; weekly during radiotherapy(until 7 weeks); 1, 2, 3 months after the end of radiotherapy
  Time from the first day of radiotherapy to the first determination of OM.
The duration of any-grade oral mucositis (OM) | 1 week before radiotherapy; weekly during radiotherapy(until 7 weeks); 1, 2, 3 months after the end of radiotherapy
  The first determination of OM to the first instance of non-OM, without a subsequent instance of OM.

OTHER OUTCOMES:
Changes of oral flora | 1 week before radiotherapy; at the middle of radiotherapy(3 weeks after the start of radiotherapy); at the end of radiotherapy(the last radiation dose received, usually 6 or 6.5 weeks).
  The changes of oral flora in patients' salivary or oral swab measured by 16s rDNA technique
Xerostomia | 1 week before radiotherapy; at the middle of radiotherapy(3 weeks after the start of radiotherapy); at the end of radiotherapy(the last radiation dose received, usually 6 or 6.5 weeks); 1, 2, 3 months after the end of radiotherapy
  Patients self-evaluated xerostomia according to Xerostomia questionnaire(score 0-100);Higher score indicates more severe symptoms
Quality of Life assessed by EORTC QLQ-C30 | 1 week before radiotherapy; at the middle of radiotherapy(3 weeks after the start of radiotherapy); at the end of radiotherapy(the last radiation dose received, usually 6 or 6.5 weeks); 1, 2, 3 months after the end of radiotherapy
  Quality of Life is assessed by EORTC QLQ-C30(European Organization for Research and Treatment of Cancer Quality of Life Questionnaire);transformed into 0-100 scales for different domains and symptoms;Higher domain scores represent better quality of life, while higher symptom scores represent worse quality of life
Quality of Life assessed by QLQ-H&N35 | 1 week before radiotherapy; at the middle of radiotherapy(3 weeks after the start of radiotherapy); at the end of radiotherapy(the last radiation dose received, usually 6 or 6.5 weeks); 1, 2, 3 months after the end of radiotherapy
  Quality of Life is assessed by QLQ-H&N35(Head and neck cancer-related quality of life scale);transformed into 0-100 scales for different domains and symptoms;Higher scores represent worse quality of life
Dysphagia | 1 week before radiotherapy; at the middle of radiotherapy(3 weeks after the start of radiotherapy); at the end of radiotherapy(the last radiation dose received, usually 6 or 6.5 weeks); 1, 2, 3 months after the end of radiotherapy
  Dysphagia is assessed by M.D.Anderson Dysphagia Inventory(score 20-100);Lower score indicates more severe symptoms
The number of dental specialist visits | The time period is the period from the start of radiotherapy to the completion of radiotherapy (usuallly 6 or 6.5 weeks).
  The number of dental specialist visits during radiotherapy between two groups
Oral health status | 1 week before radiotherapy; at the middle of radiotherapy(3 weeks after the start of radiotherapy); at the end of radiotherapy(the last radiation dose received, usually 6 or 6.5 weeks); 1, 2, 3months after the end of radiotherapy
  Oral health status encompasses several key variables: the number of natural teeth, teeth with caries, periodontal pockets, gingival bleeding, clinical attachment loss, plaque index (mean ± SD), and limited mouth opening (abnormal).
Radiotherapy interruption rate | 1 week before radiotherapy; at the middle of radiotherapy(3 weeks after the start of radiotherapy); at the end of radiotherapy(the last radiation dose received, usually 6 or 6.5 weeks).
  The number of patients who missed five or more consecutive radiations and the reasons for this are recorded during radiotherapy.

CONTACTS AND LOCATIONS:
Locations (1):
- West China Hospital, Sichuan University, Chengdu, Sichuan, China